CLINICAL TRIAL: NCT01290341
Title: A Phase 3 Double-Blind, Randomized, Placebo-Controlled,Multicenter, Parallel Group Evaluation of the Efficacy and Safety of NAFT-600 in Subjects With Tinea Pedis
Brief Title: Evaluation of the Efficacy and Safety of NAFT-600 in Subjects With Tinea Pedis
Acronym: NAFT-600
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merz North America, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MRZ 90200/3016/1
Record Dates: First submitted 2011-01-28; First posted 2011-02-07 (Estimated); Results first posted 2013-09-26 (Estimated); Last update posted 2013-09-26 (Estimated); Status verified 2013-07

CONDITIONS: Tinea Pedis
Keywords: fungal infection; athlete foot
MeSH Terms: conditions — Tinea Pedis; Mycoses | interventions — naftifine; Gels

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- NAFT-600 ( naftin 2 % gel) (Experimental): Topical; applied once daily for two weeks
  Interventions: Drug: NAFT-600 (naftin 2 % gel)
- Placebo (Placebo Comparator): Topical; applied once daily for two weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: NAFT-600 (naftin 2 % gel) — Topical; applied once daily for two weeks
  Other Names: Naftin®
  Arms: NAFT-600 ( naftin 2 % gel)
Drug: Placebo — Topical; applied once daily for two weeks.
  Arms: Placebo

SUMMARY:
This is a 6-week, double-blind, randomized, placebo-controlled, multicenter, parallel group Phase 3 study of NAFT-600 applied once a day for 2 weeks compared to vehicle (placebo) in the treatment of tinea pedis.

DETAILED DESCRIPTION:
This study is open to males and non-pregnant females, 12 years of age and over, with clinical signs and symptoms of tinea pedis consisting of at least moderate erythema, moderate scaling, mild pruritus, a positive screening KOH, and a positive culture.Subjects will be evaluated at Day 1 (baseline), Week 2, Week 4, and Week 6 (follow-up). Adverse events, concomitant medications,and study drug compliance will be reviewed at each visit. Efficacy assessments will include KOH and culture evaluations, clinical signs/symptoms (erythema, scaling, pruritus), and Investigator's Global Assessment.

ELIGIBILITY:
Inclusion Criteria:

* Males or non-pregnant females, ≥12 years of age, of any race or sex. Females of child-bearing potential must have a negative urine pregnancy test.
* For minors (less than 18 years), the parent/legal guardian must complete the informed consent process AND the subject must complete the assent process and sign the appropriate form (if age appropriate).
* Presence of interdigital only or both interdigital and moccasin types of tinea pedis on one or both feet characterized by clinical evidence of a tinea infection (at least moderate erythema, moderate scaling and mild pruritus) based on signs and symptoms in the affected area(s).

Exclusion Criteria:

* Subjects with life-threatening condition (ex. autoimmune deficiency syndrome, cancer, unstable angina or myocardial infarction) within the last 6 months.
* Subjects with abnormal findings - physical or laboratory - that are considered by the investigator to be clinically important and indicative of conditions that might complicate interpretation of study results.
* Subjects with a known hypersensitivity to study drugs or their components.
* Subjects who have a recent history or who are currently known to abuse alcohol or drugs.
* Uncontrolled diabetes mellitus.
* Hemodialysis or chronic ambulatory peritoneal dialysis therapy.
* Current diagnosis of immunocompromising conditions.
* Foot psoriasis, corns and/or callus involving any web spaces, atopic or contact dermatitis.
* Severe dermatophytoses, onychomycosis (on the evaluated foot), mucocutaneous candidiasis or bacterial skin infection.
* Extremely severe tinea pedis (incapacitating).
* Female subject who is pregnant or lactating, who is not using or does not agree to use an acceptable form of contraception during the study, or who intends to become pregnant during the study.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 860 (Actual)
Dates: Start 2011-02; Primary Completion 2011-11 (Actual); Study Completion 2011-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lawrency Parrish, MD, Principal Investigator — Paddington Testing Co., Inc.
Locations (23):
- United States (23):
  - Radiant Research, Inc., Tucson, Arizona
  - T. Joseph Raoof, MD, Inc., Encino, California
  - Walter K. Nahm, MD, PhD, Inc., San Diego, California
  - Colorado Medical Research Center, Denver, Colorado
  - Longmont Clinic, PC, Longmont, Colorado
  - Tampa Bay Medical Research, Clearwater, Florida
  - Lake Washington Foot and Ankle Center, Melbourne, Florida
  - Clinical Research Atlanta, Stockbridge, Georgia
  - Hudson Dermatology, Evansville, Indiana
  - Department of Veterans Affairs, Minneapolis, Minnesota
  - Academic Dermatology Associates, Albuquerque, New Mexico
  - Radiant Research, Inc, Cincinnati, Ohio
  - Radiant Research, Inc., Columbus, Ohio
  - Oregon Dermatology & Research Center, Portland, Oregon
  - Temple University- School of Podiatric Medicine, Philadelphia, Pennsylvania
  - Palmetto Clinical Trial Services, LLC, Simpsonville, South Carolina
  - DermResearch, Inc., Austin, Texas
  - J&S Studies, Inc., College Station, Texas
  - Research Across America, Dallas, Texas
  - Endeavor Clinical Trials, PA, San Antonio, Texas
  - Progressive Clinical Research, San Antonio, Texas
  - The Education and Research Foundation, Inc., Lynchburg, Virginia
  - Madison Skin and Research, Inc, Madison, Wisconsin

RESULTS

PARTICIPANT FLOW:
Groups:
- NAFT-600; Placebo: Topical; applied once daily for two weeks
Period: Overall Study
Arm/Group | NAFT-600 | Placebo
Started | 573 | 287
Completed | 481 | 258
Not Completed | 92 | 29
Not completed — Protocol Violation | 7 | 3
Not completed — Adverse Event | 1 | 0
Not completed — Lost to Follow-up | 21 | 10
Not completed — Withdrawal by Subject | 19 | 5
Not completed — Negative baseline culture and others | 44 | 11

BASELINE CHARACTERISTICS:
Population: The Safety Evaluation Set (SES) which is the population of subjects who receive at least one dose of study medication is used.
Groups:
- Total: Total of all reporting groups
Arm/Group | NAFT-600 | Placebo | Total
Number analyzed (Participants) | 572 | 287 | 859
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 15 | 4 | 19
  Between 18 and 65 years | 500 | 252 | 752
  >=65 years | 57 | 31 | 88
Age Continuous [Mean (Standard Deviation); unit: years] | 45.2 (14.9) | 45.2 (14.7) | 45.2 (14.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 118 | 73 | 191
  Male | 454 | 214 | 668
Region of Enrollment [Number; unit: participants]
  United States | 572 | 287 | 859

OUTCOME MEASURES:

1. Primary Outcome: Complete Cure of Interdigital Tinea Pedis
Description: The primary efficacy comparison between NAFT-600 gel and placebo will be based on the percentage of subjects at Week 6 with complete cure of interdigital tinea pedis.
  Complete cure is defined as negative mycology results (dermatophyte culture and KOH) and the absence of erythema, scaling, and pruritus.
Time Frame: Visit 4/ Week 6
Population: Full Analysis Set (FAS) defined as the subset of all subjects in the Safety Evaluation Set (SES) with a positive mycology culture at baseline and for whom the primary efficacy variable is available. This was a modified intent to treat principle because the culture results were not available before the start of treatment.
Measure: Number; unit: percentage of subjects
Arm/Group | NAFT-600 | Placebo
Number analyzed (Participants) | 400 | 213
percentage of subjects | 26.0 | 3.3
Statistical Analysis 1: Comparison: NAFT-600 vs Placebo; In order to compare complete cure rate in the NAFT-600 group with that of the Placebo group, the following one-sided hypothesis test was carried out: H0 (null): p1<=p0 versus Ha (alternate): p1>p0, where p0 and p1 are the proportions of subjects with complete cure in the placebo and NAFT-600 treatment groups respectively; Test type: Superiority or Other; p < 0.025, Cochran-Mantel-Haenszel; The CMH test statistic after stratification by site was used to compare subjects with complete cure between NAFT-600 and Placebo; p-value = 0.001

2. Secondary Outcome: Effective Treatment and Mycological Cure of Interdigital Tinea Pedis at Week 6
Description: Effective treatment of interdigital tinea pedis which is defined as negative KOH and negative dermatophyte culture and erythema, scaling, and pruritus scores of 0 or 1 (corresponding to absent and mild respectively).
  Mycological cure of interdigital tinea pedis which is defined as negative KOH and negative dermatophyte culture.
Time Frame: Visit 4/ Week 6
Population: Full Analysis Set (FAS) using a Modified Intent to Treat (MITT) population.
Measure: Number; unit: percentage of subjects
Arm/Group | NAFT-600 | Placebo
Number analyzed (Participants) | 400 | 213
percentage of subjects
  Mycological Cure | 58.8 | 10.3
  Effective Treatment | 50.8 | 7.0

ADVERSE EVENTS:
Time Frame: Adverse Events were collected up to Week 6.
Arm/Group | NAFT-600 | Placebo
Serious Adverse Events (participants affected / at risk) | 1/572 | 2/287
Other Adverse Events (participants affected / at risk) | 16/572 | 5/287
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | NAFT-600 (N=572) | Placebo (N=287)
Urethral Stenosis (Renal and urinary disorders) | 1 | 0
Appendicitis (Infections and infestations) | 0 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | NAFT-600 (N=572) | Placebo (N=287)
Headache (Nervous system disorders) | 16 | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Institution and Principal Investigator agreed not to individually publish or assist other person or entity with any articles, papers, and/or make presentations, speeches referring to the protocol, clinical trial data, the study, or the study drug or any data, results, materials, or information generated or obtained by the Institution or the Principal Investigator without the prior written consent of Merz, which consent may be withheld in the sole discretion of Merz.